CLINICAL TRIAL: NCT01410630
Title: FLT-PET/CT vs FDG-PET/CT for Therapy Monitoring of Diffuse Large B-cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-001275; SU-07072011-8046 (Other: Stanford University); 19997 (Other: Stanford IRB); 17-001275 (Other: UCLA IRB); JCCCID811 (Other: Jonsson CCC)
Record Dates: First submitted 2011-07-22; First posted 2011-08-05 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma; Lymphoma, Non-Hodgkin; Large B Cell Diffuse Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FLT-PET/CT and FDG-PET/CT scan: Patients will have FLT-PET/CT and FDG-PET/CT scans performed 18-24 days after the second cycle of R-CHOP.
  Interventions: Diagnostic Test: FLT-PET/CT; Diagnostic Test: FDG-PET/CT; Drug: FLT

INTERVENTIONS:
Diagnostic Test: FLT-PET/CT — Standard of Care
  Other Names: FLT Positive Emission Tomography
Diagnostic Test: FDG-PET/CT — Standard of Care
  Other Names: FDB Positive Emission Tomography
Drug: FLT — 5 mCi IV
  Other Names: fluoro-L-thymidine

SUMMARY:
A research study of a new method of visualizing internal organs called 18F-FLT PET/CT that yields better tracking of cancer treatment progress. PET/CT stands for positron emission tomography with low dose computed tomography and has been used for many years. 18F-FLT PET/CT uses a new tracer, fluorothymidine, which is taken up by cells that are actively proliferating or dividing such as cancer cells. We hope to learn whether this tracer is superior to the conventional tracer for monitoring treatment of diffuse large B-cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
-Primary Objective

Investigate whether the PPV of FLT-PET/CT is significantly higher than that of FDG-PET/CT by following up patients for at least 24 months post-therapy or until evidence of persistent disease/disease progression.

-Secondary Objectives

Investigate whether the event free survival (EFS) of patients with FDG-PET/CT-positive and FLT-PET/CT negative scans is not significantly lower than that of patients with concordantly negative FDG-PET/CT and FLT-PET/CT scans and that the NPV or FLT-PET/CT is similar to that of FDG-PET/CT

Correlate interim FLT-PET/CT and FDG-PET/CT with the International Prognostic Index (IPI), a well-established predictor of outcome in DLBCL, to determine their independent prognostic value from the IPI

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a histologic or cytological diagnosis of de novo DLBCL and be scheduled to receive first line chemotherapy with R-CHOP given every 21 days (R-CHOP-21) within 6 weeks of their enrollment and for 6 cycles.
* Patients must be >=18 years of age, but there will be no discrimination based on gender, race, creed, or ethnic background.
* Patients must have an ECOG performance status of 0-2.
* Patients must sign an informed consent, and be mentally responsible.

Exclusion Criteria:

* Subjects with significant concurrent medical complications that in the judgment of the Principal Investigator(s) could affect the patient's ability to complete the planned trial, including the multiple imaging studies.
* Patients with history of prior lymphoma (e.g., follicular lymphoma) and/or second cancers other than basal cell carcinoma.
* Patients planned to be treated with R-CHOP-14 (i.e., R-CHOP given every 14 days) will be excluded (this should be extremely rare, if at all, since R-CHOP-21 is the standard treatment.
* Patients who are scheduled to receive Rituxan or any other therapy (e.g., XRT, radioimmunotherapy) as adjuvant therapy after completion of R-CHOP-21.
* Pregnant women will be excluded.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) after study entry and for the duration of study participation. The effects of FLT on the developing human fetus are unknown. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A screening urine human chorionic gonadtropin (hCG) (pregnancy test) will be administered in Nuclear Medicine to women of childbearing potential before each FLT scan and pregnant women will be stopped from participating further in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 18 years of age or older
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) of 3'-deoxy-3'-[F-18]-fluorothymidine (FLT) Positron emission tomography (PET/CT) versus Fluorodeoxyglucose (FDG)PET/CT | 24 Months

SECONDARY OUTCOMES:
Overall survival after initiation of therapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Quon, MD, Principal Investigator — University of California at Los Angeles
Locations (4):
- United States (3):
  - University of California at Los Angeles, Los Angeles, California
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
- Aachen University, Aachen, Germany